CLINICAL TRIAL: NCT03317990
Title: A Single Blinded, IDEAL Stage 3, Multi-Centre, Randomised Controlled Trial to Assess NeuroSAFE Robotic Assisted Radical Prostatectomy (RARP) vs Standard Robotic Assisted Radical Prostatectomy (RARP) in Men With Prostate Cancer
Brief Title: Evaluating the Effects of Frozen Section Technology on Oncological and Functional Outcomes at Radical Prostatectomy.
Acronym: NeuroSAFEPROOF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: North Bristol NHS Trust (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); University College London Hospitals (Other); NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 220262; 17/0443 (Other Grant/Funding Number: University College London)
Record Dates: First submitted 2017-10-05; First posted 2017-10-23 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Nerve sparing; NeuroSAFE; Frozen section
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: A single blinded, multi-centre, randomised controlled trial. Parallel group, two-arm, with 1:1 allocation ratio between nerve sparing guided by NeuroSAFE and current UK practice (guided by MRI, biopsy and clinical examination).
Who Masked: Participant
Masking Description: Patients will be blinded as to whether the person has had NeuroSAFE procedure. The surgeon and pathologist cannot be blinded to this.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NeuroSAFE procedure (Experimental): These patients will undergo robotic radical prostatectomy with bilateral nerve spare.The pathologist will remove the pre-painted surface of the gland (which had been in contact with the neurovascular bundles) using a sharp blade.The tissue sample will be snap frozen and embedded in OCT.Using a cryostat, 10 micron thick slices will be placed on slides.The entire length of the area of interest will be sampled in this way generating ≈10 frozen sections per side.The slides will be stained with H&E and will be examined by a consultant pathologist.As soon as examination is complete the pathologist will telephone the operating surgeon to give the result.Presence of cancer cells at the margin of resection constitutes a positive margin and the neurovascular bundle on that side will be resected if the PSM is present in more than one slice on the same side or for a distance of 3 or more mm.
  Interventions: Procedure: NeuroSAFE procedure
- Control (Active Comparator): These patients will undergo robotic radical prostatectomy with a nerve sparing procedure based on surgical planning performed by a consultant radiologist. The mp-MRI will be reviewed by a consultant radiologist along with the details of the prostate biopsy and DRE a decision to perform unilateral, bilateral or non-nerve sparing will be established and recorded in the clinical record form (CRF) for each patient.
  Interventions: Procedure: Standard RARP

INTERVENTIONS:
Procedure: NeuroSAFE procedure — When the prostate is removed from within the patient as it is disconnected from its attachments. The specimen will then be painted (right=blue, left =black) by the operating surgeon and delivered expediently to the pathologist who will perform frozen section analysis of the painted areas. The pathologist will remove the pre-painted surface of the gland (which had been in contact with the neurovascular bundles) using a sharp blade. The tissue sample will be snap frozen and embedded in OCT. If a significant positive margin (on more than one section from one side or in a single section but greater than or equal to 3mm) is reported by the pathologist, the entire neurovascular bundle on the affected side will be removed and sent for formal pathological examination.
  Other Names: NeuroSAFE RARP
  Arms: NeuroSAFE procedure
Procedure: Standard RARP — Patients will undergo the standard intervention - RARP without NeuroSAFE Frozen section analysis
  Arms: Control

SUMMARY:
In summary this trial will test whether this new surgical technique can be used to make surgery safer and more effective whilst allowing improved quality of life for patients having surgery for prostate cancer. If the technique is proven effective the investigators will use the experience gained to promote its use throughout the NHS through training courses and publication and dissemination of the resultant data. Staff from centres participating in this trial will be fully trained in the NeuroSAFE technique.

A patient and public involvement afternoon was held for participants of the NeuroSAFE PROOF feasibility study, family members, men with prostate cancer, and staff members at UCLH. The event was supported by the charity Orchid Cancer appeal. The high levels of attendance was demonstrative of the support within our patient group for the work of this trial. The trial team listened to the comments made by participants and members of the public and have made some changes to the design of our trial as a result of this feedback.

DETAILED DESCRIPTION:
Prostate cancer is very common and results in the death of many men in the developed world. Prostate cancer that has not spread outside the prostate can usually be cured by surgical removal of the prostate gland (radical prostatectomy).

Radical Prostatectomy can be associated with urinary incontinence due to damage to the involuntary sphincter and erectile dysfunction due to damage of the nerves that run within the outer coverings of the prostate. Surgical sparing of these nerves to preserve quality of life may risk leaving cancer cells behind often meaning that the patients need extra treatment with radiotherapy. This trial is designed to evaluate a new method designed to decrease the risk of compromising cancer control associated with sparing of the nerves as well as evaluate effects on the need for radiotherapy after surgery if cancer is left behind. The Investigators will also evaluate effects on the quality of life in patients who have undergone RARP. The trial is needed now because the nature of prostate cancers treated surgically is changing rapidly. The techniques developed in low risk cancer to spare the nerves which run alongside the prostate, may not necessarily be safe when used on the more aggressive cancers operated on nowadays and if they are adopted without adequate investigation, the risk is that patients will be exposed to increased risk of cancer recurrence and needing extra treatment with radiotherapy with consequent side effects and extra cost to the NHS.

On the outside of the prostate, within its outermost coverings, run the nerves thought to be responsible for producing erections. Preservation of these nerves has also been linked to more rapid reestablishment of urinary continence following surgical removal of the prostate. Robotic technology has been developed which allows the prostate to be removed through very small incisions. The surgeons view is magnified in 3D, which facilitates the peeling off of the outer layers, containing the nerves (so called nerve sparing). With nerve sparing the nerves controlling erections are left intact whilst the prostate itself, along with the cancer within it, is removed.

This increases the patient's chances of getting erections of sufficient quality for penetrative sex. Data from several case series, including our own, suggest that the higher the degree of nerve sparing performed, the more likely a patient is to be potent and continent of urine. In our series, bilateral nerve sparing results in 85% of men being able to get usable erections*, whereas only 45% of men will have useable erections* when only one side is spared.

Nerve sparing has largely been developed and the effects have been evaluated in the USA where prostate cancer is detected at an earlier stage because PSA screening is performed commonly. In the UK, where PSA screening is not commonly carried out, tumours resected at surgery are larger and more aggressive, often having spread through the capsule of the prostate. In addition, the move away from surgery for small low-grade tumours in the UK means that the prostate cancers treated by surgery are larger and more aggressive overall. This means that the tumours are closer to the outer limit of the prostate because the more aggressive tumours tend to work their way out through the outer capsule of the prostate. A nerve sparing approach is associated with an increased risk that tumour will be left on the surface of the resected specimen. This is referred to as a positive surgical margin (PSM). One of the principles of (radical) cancer surgery is that cancerous tissue should be removed with a covering of non-cancerous tissue to give the best chance of cure (a so called negative or clear surgical margin). Positive surgical margins are associated with an increased chance of recurrence following surgery and require further treatment, usually with radiotherapy, which is expensive and engenders its own side effects. The investigators plan to evaluate the use of a modified version of a frozen section technique called NeuroSAFE in promoting nerve sparing without diminishing the oncological effects of surgery by generating PSMs. During this frozen section technique, once the prostate is removed, the areas of prostate adjacent to the spared nerves are sliced from the surgical specimen and rapidly frozen and stained so that they can be examined carefully by a pathologist. If the pathologist identifies a significant positive surgical margin, the spared nervous tissue on that side will be surgically resected before the patient is woken up at the end of the operation. When this is done the cancer behaves as if it had been resected with a negative surgical margin at the outset. Frozen section analysis does not add much time to the surgical procedure, as once the prostate is removed, the rest of the operation (joining the bladder to the urethra and removing pelvic lymph nodes) can proceed whilst the frozen section analysis is performed. Patients enrolled to the trial will be randomised between A) standard UK nerve sparing practice, wherein the degree to which the nerves can be spared is determined by the operating surgeon based on clinical examination, biopsy results and multi-parametric MRI and B) bilateral nerve sparing with frozen section analysis.

The Trial team recently surveyed UK robotic prostatectomists and confirm that currently UK surgeons predominately rely on MRI, biopsy and Digital Rectal Exam (DRE) findings to determine whether they can spare nerves, but that there is little consistency in the means by which a surgeon decides whether or not they can spare nerves in a particular case. Our survey tells us that UK surgeons do not use frozen section to direct nerve sparing with only 5% of UK prostatectomists ever having used it at all.

What are the potential outcomes of this research? This trial will provide a thorough evaluation of a new technique designed to minimise the occurrence of PSM and exposure to extra treatment or cancer recurrence. It will generate vital data regarding the cost/benefit of using this procedure. The relationship between the degree and frequency of nerve sparing on quality of life will be evaluated in terms of sexual potency and urinary continence in UK patients undergoing RALP. The assessment of these functions will include patient reported outcomes.

* At 2 years following surgery using Viagra or an equivalent PDE5i.

ELIGIBILITY:
Inclusion Criteria:

1. Men opting to undergo RARP for organ confined prostate cancer.
2. Potent men (IIEF 22-25 not using PDE5i or other medications or vacuum pump)
3. Men who are continent of urine (no self-reported urinary incontinence)
4. Has given written informed consent
5. Ability to read English sufficiently to answer questionnaires and understand PIS

Exclusion Criteria:

1. Unable to undergo robotic prostatectomy
2. Known urinary incontinence
3. Previous treatment for prostate cancer
4. Previous/current hormone treatment for prostate cancer
5. Nerve sparing deemed futile due to locally advanced disease by surgeon and radiologist

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2027-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Greg L Shaw, MD, Principal Investigator — University College, London
Locations (5):
- United Kingdom (5):
  - North Bristol NHS Trust, Bristol
  - NHS Greater Glasgow & Clyde, Glasgow
  - University College London Hospital, London
  - Nottingham University Hospitals, Nottingham
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Once primary outcome data is published, a limited, pseudonymised dataset for the primary outcomes that underlie the results reported in the final manuscript along with the data dictionary will be available to be shared. All data (pseudonymised) will remain under the custodianship of the trial management group (TMG). Requests for data are submitted to the committee via (ncita.neurosafe@ucl.ac.uk). A data access agreement will need to be signed. As the NeuroSAFE PROOF study is ongoing, we will not share the full dataset until follow-up of participants is completed and the long-term follow up final manuscript has been published.
Supporting Information: Study Protocol
Time Frame: Once primary outcome data is published in the final manuscript
Access Criteria: A limited, pseudonymised dataset for the primary outcomes that underlie the results reported in the final manuscript along with the data dictionary will be available to be shared. All data (pseudonymised) will remain under the custodianship of the trial management group (TMG). Requests for data are submitted to the committee via (ncita.neurosafe@ucl.ac.uk). A data access agreement will need to be signed. As the NeuroSAFE PROOF study is ongoing, we will not share the full dataset until follow-up of participants is completed and the long-term follow up final manuscript has been published.
URL: https://pubmed.ncbi.nlm.nih.gov/35869497/

REFERENCES:
- [Background] https://doi.org/10.6084/m9.figshare.27054979.v1
- [Background] Beyer B, Schlomm T, Tennstedt P, Boehm K, Adam M, Schiffmann J, Sauter G, Wittmer C, Steuber T, Graefen M, Huland H, Haese A. A feasible and time-efficient adaptation of NeuroSAFE for da Vinci robot-assisted radical prostatectomy. Eur Urol. 2014 Jul;66(1):138-44. doi: 10.1016/j.eururo.2013.12.014. Epub 2013 Dec 24. PMID 24411279
- [Background] Vasdev N, Agarwal S, Rai BP, Soosainathan A, Shaw G, Chang S, Prasad V, Mohan-S G, Adshead JM. Intraoperative Frozen Section of the Prostate Reduces the Risk of Positive Margin Whilst Ensuring Nerve Sparing in Patients with Intermediate and High-Risk Prostate Cancer Undergoing Robotic Radical Prostatectomy: First Reported UK Series. Curr Urol. 2016 May;9(2):93-103. doi: 10.1159/000442860. Epub 2016 May 20. PMID 27390582
- [Derived] Dinneen E, Almeida-Magana R, Al-Hammouri T, Pan S, Leurent B, Haider A, Freeman A, Roberts N, Brew-Graves C, Grierson J, Clow R, Williams N, Aning J, Walton T, Persad R, Oakley N, Ahmad I, Dutto L, Briggs T, Allen C, Tandogdu Z, Adshead J, Oxley J, Kelly J, Shaw G; NeuroSAFE PROOF Investigators. Effect of NeuroSAFE-guided RARP versus standard RARP on erectile function and urinary continence in patients with localised prostate cancer (NeuroSAFE PROOF): a multicentre, patient-blinded, randomised, controlled phase 3 trial. Lancet Oncol. 2025 Apr;26(4):447-458. doi: 10.1016/S1470-2045(25)00091-9. Epub 2025 Mar 24. PMID 40147459
- [Derived] Dinneen E, Grierson J, Almeida-Magana R, Clow R, Haider A, Allen C, Heffernan-Ho D, Freeman A, Briggs T, Nathan S, Mallett S, Brew-Graves C, Muirhead N, Williams NR, Pizzo E, Persad R, Aning J, Johnson L, Oxley J, Oakley N, Morgan S, Tahir F, Ahmad I, Dutto L, Salmond JM, Kelkar A, Kelly J, Shaw G. NeuroSAFE PROOF: study protocol for a single-blinded, IDEAL stage 3, multi-centre, randomised controlled trial of NeuroSAFE robotic-assisted radical prostatectomy versus standard robotic-assisted radical prostatectomy in men with localized prostate cancer. Trials. 2022 Jul 22;23(1):584. doi: 10.1186/s13063-022-06421-7. PMID 35869497
- [Derived] Almeida-Magana R, Maroof H, Grierson J, Clow R, Dinneen E, Al-Hammouri T, Muirhead N, Brew-Graves C, Kelly J, Shaw G. E-Consent-a guide to maintain recruitment in clinical trials during the COVID-19 pandemic. Trials. 2022 May 12;23(1):388. doi: 10.1186/s13063-022-06333-6. PMID 35550639
- [Derived] Dinneen E, Haider A, Grierson J, Freeman A, Oxley J, Briggs T, Nathan S, Williams NR, Brew-Graves C, Persad R, Aning J, Jameson C, Ratynska M, Ben-Salha I, Ball R, Clow R, Allen C, Heffernan-Ho D, Kelly J, Shaw G. NeuroSAFE frozen section during robot-assisted radical prostatectomy: peri-operative and histopathological outcomes from the NeuroSAFE PROOF feasibility randomized controlled trial. BJU Int. 2021 Jun;127(6):676-686. doi: 10.1111/bju.15256. Epub 2021 Mar 29. PMID 32985121
- [Derived] Dinneen E, Haider A, Allen C, Freeman A, Briggs T, Nathan S, Brew-Graves C, Grierson J, Williams NR, Persad R, Oakley N, Adshead JM, Huland H, Haese A, Shaw G. NeuroSAFE robot-assisted laparoscopic prostatectomy versus standard robot-assisted laparoscopic prostatectomy for men with localised prostate cancer (NeuroSAFE PROOF): protocol for a randomised controlled feasibility study. BMJ Open. 2019 Jun 11;9(6):e028132. doi: 10.1136/bmjopen-2018-028132. PMID 31189680

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 364 evaluable participants were required to have 80% power to detect such difference, with a two-sided α of 5%. Allowing for a 10% dropout rate, we aimed to recruit 404 participants (202 per group).
Pre-assignment Details: A total of 364 evaluable participants were required to have 80% power to detect such difference, with a two-sided α of 5%. Allowing for a 10% dropout rate, we aimed to recruit 404 participants (202 per group).
Period: Overall Study
Arm/Group | NeuroSAFE Procedure | Control
Started | 204 | 203
Patients Who Underwent Surgery | 190 | 191
Completed | 174 | 173
Not Completed | 30 | 30

BASELINE CHARACTERISTICS:
Population: Patients who underwent surgery
Groups:
- Total: Total of all reporting groups
Arm/Group | NeuroSAFE Procedure | Control | Total
Number analyzed (Participants) | 190 | 191 | 381
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.8 (6.4) | 57.3 (7) | 57.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 190 | 191 | 381
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity data was self-reported following the England and Wales 2021 census categories Population: Only patient with known race/ethnicity data were included, the rest have missing data
  Participants
    Ethnicity: number analyzed (Participants) | 171 | 169 | 340
    Ethnicity: White | 108 | 103 | 211
    Ethnicity: Black | 49 | 53 | 102
    Ethnicity: Asian | 9 | 9 | 18
    Ethnicity: Other/Mixed | 5 | 4 | 9
Baseline PSA [Mean (Standard Deviation); unit: Ng/ml] — Population: Only patient with known BMI data were included, the rest have missing data
  Ng/ml
    number analyzed (Participants) | 188 | 191 | 379
    (all) | 9.1 (6.5) | 8.6 (5.9) | 8.9 (6.2)
Clinical T-Stage [Count of Participants; unit: Participants] — Clinical T staging based on TNM Staging Categories before surgery T1 The tumour is not detectable by physical examination or imaging T2 The tumour appears confined to the prostate T3 The tumour has features suggestive of extracapsular extension Population: Only patients with known T staging classification were included, rest have missing data
  Participants
    number analyzed (Participants) | 180 | 179 | 359
    T-1 | 7 | 6 | 13
    T-2 | 135 | 132 | 267
    T-3 | 38 | 41 | 79
Cambridge Prognostic Group [Count of Participants; unit: Participants] — The Cambridge Prognostic Group (CPG) classification is a five-tiered system used to predict prostate cancer progression and mortality. This system categorizes patients into groups based on three factors at the time of diagnosis: PSA levels, Gleason Grade Group from the biopsy, and clinical T staging. Group 1 represents the lowest risk of prostate cancer specific mortality and Group 5 the highest. Population: Only patients with complete staging information were included in this analysis
  Participants
    number analyzed (Participants) | 177 | 179 | 356
    1 | 6 | 4 | 10
    2 | 80 | 83 | 163
    3 | 38 | 40 | 78
    4 | 46 | 44 | 90
    5 | 7 | 8 | 15
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body mass index
  kg/m^2 | 27.3 (3.8) | 27.1 (3.4) | 27.2 (3.6)
Baseline IIEF-5 Score [Mean (Standard Deviation); unit: units on a scale] — The International Index of Erectile Function-5 (IIEF-5) measures erectile dysfunction severity. Total scores range from 5 to 25, calculated by summing 5 items. Higher scores indicate better erectile function. Severity categories: 22-25 = no erectile disfunction, 17-21 = mild, 12-16 = mild to moderate, 8-11 = moderate, 5-7 = severe. No subscales are used; the total score is the sum of all items.
  units on a scale | 23.3 (2.2) | 23.3 (2.5) | 23.3 (2.4)
Prostate volume [Mean (Standard Deviation); unit: cm^3] | 38.1 (17.6) | 39.7 (20.1) | 38.9 (18.9)

OUTCOME MEASURES:

1. Primary Outcome: Erectile Function
Description: Comparison of the erectile function at 12-months according to allocated treatment arm (i.e. NeuroSAFE RARP [intervention] vs. standard RARP [control]). Erectile function is measured using the IIEF-5 questionnaire
  Measure Description: The International Index of Erectile Function-5 (IIEF-5) measures erectile dysfunction severity. Total scores range from 5 to 25, calculated by summing 5 items. Higher scores indicate better erectile function. Severity categories: 22-25 = no erectile disfunction, 17-21 = mild, 12-16 = mild to moderate, 8-11 = moderate, 5-7 = severe. No subscales are used; the total score is the sum of all items.
Time Frame: 1 year
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NeuroSAFE Procedure | Control
Number analyzed (Participants) | 173 | 171
units on a scale | 12.7 (8.0) | 9.7 (7.5)
Statistical Analysis 1: Comparison: NeuroSAFE Procedure vs Control; Normal linear regression model adjusted for recruitment site, participant's age, and IIEF-5 at baseline, in participants with available data; Test type: Superiority; p < 0.0001, Regression, Linear; Mean Difference (Final Values) = 3.18, 95% CI 2-sided [1.62 to 4.75]

2. Secondary Outcome: Functional Outcome - Urinary Continence
Description: Comparison of the continence at 3 months, measured using the ICIQ questionnaire between intervention and control arms.
  o Additional subgroup analysis: restricted to men who did not receive a pre-operative radiologist recommendation for bilateral nerve sparing
  The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) assesses the frequency, severity, and impact of urinary incontinence. Total scores range from 0 to 21, with higher scores indicating more severe symptoms. Scores are calculated by summing 3 scored items. No subscales are used; higher values represent worse outcomes.
Time Frame: 3 months
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NeuroSAFE Procedure | Control
Number analyzed (Participants) | 158 | 158
units on a scale | 5.8 (4.1) | 7.4 (5.2)
Statistical Analysis 1: Comparison: NeuroSAFE Procedure vs Control; Test type: Superiority; p = 0.006, Regression, Linear; Mean Difference (Final Values) = -1.41, 95% CI 2-sided [-2.42 to -0.41]

3. Secondary Outcome: Functional Outcome - Urinary Continence at 6 Months
Description: as for outcome 2
Time Frame: 6 months
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NeuroSAFE Procedure | Control
Number analyzed (Participants) | 145 | 158
units on a scale | 4.5 (4.2) | 5.1 (4.7)

4. Secondary Outcome: Oncological Outcome
Description: Oncological outcome will be classified into four categories according to the following definition:
  1. PSA persistence : PSA≥0.2 at visit 2
  2. Biochemical recurrence: (PSA less than 0.2 at visit 2) and (PSA≥0.2 at visit 3 or PSA≥0.2 at visit 4)
  3. Early salvage treatment: (PSA less than 0.2 at each of visit 2, visit 3, and visit 4) and (received adjuvant treatment in the first year)
  4. Other (No recurrence or treatment): (PSA less than 0.2 at each of visit 2, visit 3, and visit 4) and did not receive adjuvant treatment
Time Frame: 12 months after surgery
Population: Participants with available data
Measure: Count of Participants; unit: Participants
Arm/Group | NeuroSAFE Procedure | Control
Number analyzed (Participants) | 182 | 188
Participants
  PSA persistance | 7 | 5
  Biochemical recurrence | 10 | 7
  Adjuvant treatment | 8 | 2
  Other (no recurrence or treatment) | 157 | 174

5. Secondary Outcome: Quality of Life - EQ-5D-5L
Description: A comparison of the proportion of men achieving the best quality of life according to the EQ-5D-5L between intervention and control arms.
Time Frame: 12 months and 24 months
Reporting Status: Not Posted

6. Secondary Outcome: Quality of Life - EQ-5D-5L Score
Description: Analysis of EQ-5D-5L scores to produce QALYs at 12 months by arm
Time Frame: 12 months and 24 months
Reporting Status: Not Posted

7. Secondary Outcome: Oncological Outcomes - Positive Surgical Margins
Description: Descriptive tabulation of PSM rates between NeuroSAFE RARP and standard RARP arms. PSMs will be grouped as:
  1. Negative surgical margins
  2. Small single positive surgical margin
  3. Large or multifocal surgical margin
Time Frame: At the time of intervention
Population: Participants with available data
Measure: Count of Participants; unit: Participants
Arm/Group | NeuroSAFE Procedure | Control
Number analyzed (Participants) | 190 | 191
Participants
  Negative | 124 | 137
  Small single positive surgical margin | 40 | 24
  >3 mm or multifocal positive surgical margin | 26 | 30

8. Secondary Outcome: Health Economic Analysis
Description: Use of the Health Economics Questionnaires to inform a health cost analysis of NeuroSAFE RARP vs. standard RARP.
  * Economic analysis to assess healthcare resources use by arm and cost analysis to assess:
  * Cost of intervention and control
  * Cost of NHS resource use (medications, physiotherapy,
  * Cost of private health care resources (medication, physiotherapy)
  * Other private/societal costs (productivity losses, caregivers costs, out of pocket cost for transport, equipment)
Time Frame: 12 months and 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From surgery to 90 postoperative days
Description: Adverse events and serious adverse events occurring within 90 days of surgery were reported descriptively, numbers reflect patients who had surgery
Arm/Group | NeuroSAFE Procedure | Control
All-Cause Mortality (participants affected / at risk) | 2/190 | 2/191
Serious Adverse Events (participants affected / at risk) | 6/190 | 5/191
Other Adverse Events (participants affected / at risk) | 0/190 | 0/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NeuroSAFE Procedure (N=190) | Control (N=191)
Postoperative haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Unrelated hospital readmission (General disorders) | 1 (1) | 0 (0)
Postoperative haemorrhage (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pelvic haematoma (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Urethro-vesical anastomosis leak (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incidental non-tension pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infected scrotal haematoma (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Several limitations are to be mentioned. First, oncological outcomes are limited to 12 months, most procedures were performed at one centre, clinical research team members who conducted the follow-up assessments were aware of treatment allocation. Definition and analysis methods for the primary outcome was changed after the study commenced.

Results analysis is ongoing; results on quality of life, health economic analysis, and 2 year functional and oncological outcomes will be published in 2026.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT03317990/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT03317990/SAP_001.pdf